CLINICAL TRIAL: NCT07359495
Title: Effect of a Multicomponent Exercise Program on Muscle Quality Assessed by Ultrasound, Body Composition, and Functionality in Older Women: A Randomized Controlled Trial Protocol
Brief Title: Multicomponent Training and Muscle Quality in Older Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Luis Polo Ferrero, Professor, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USalamancaMTUS
Record Dates: First submitted 2025-12-15; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Sarcopenia
Keywords: Healthy aging; Muscle Quality; Physical Function; Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Multicomponent training) (Experimental): Participants in this group will follow the multi-component exercise programme. The load progression will be based on individual perceived exertion. At the beginning of the intervention, participants will be taught how to interpret the modified Borg scale. At the end of each week, each person's perception of exertion will be recorded in relation to the three sessions completed. The aim will be to maintain a constant level of between 5 and 7 on the scale, which corresponds to 'hard' and 'very hard'. If the perceived exertion is greater than 7, it will be reduced, and conversely, if it is less than 5, the intensity will be increased.
  Interventions: Other: Multicomponent training
- Control Group (No Intervention): Participants in this group will maintain their usual diet and physical activity, without changing their habits during the intervention period. They will not participate in other physical exercise programs, nor will they engage in frequent and systematic physical exercise.

INTERVENTIONS:
Other: Multicomponent training — The exercise battery includes lower body work (squats, deadlifts, front and sagittal plane lunges, hip abduction/extension, and plantar flexion) and upper body work (wall flexion-extensions, shoulder raises, and elbow flexion-extensions). In addition to the strength exercises mentioned above, balance exercises such as walking in tandem, standing on one leg, side steps, and weight transfer will also be performed. Aerobic capacity will be worked on by walking at a moderate intensity, and flexibility will be improved through stretching the main muscle groups.
  Arms: Intervention Group (Multicomponent training)

SUMMARY:
This study aims to evlauate the effect os a 32-week multicomponent training (MT) program on muscle architecture and muscle quality (assessed by ultrasound) in womer over 60 years. The study will also analyze concurrent changes in muscle strength, physical performance, and body composition. The hypothesis is that the training will induce positive architectural adaptations, such as reduced echogenicity and increased thickness in the rectus femoris and rectus abdominis muscles, correlating with improved functional independence.

DETAILED DESCRIPTION:
Population aging emphasizes the need for "healthy aging", where muscle quality (MQ) is a vital metric. However, there is a lack of robust longitudinal protocols integrating ultrasound-assessed MQ with functional performance in older women. This randomized controlled trial involves community-dwelling women aged 60+ from the Geriatric Revitalization Program in Salamanca. Participants will be randomized (1:1) into an experimental group (multicomponent training) or a control group. The intervention is a 32-week supervised program (3 sessions/week, 50 min/session) combining aerobic, strength, balance, and coordination exercises. Primary outcomes focus on muscle architecture (echo intensity and thickness) in the rectus femoris and rectus abdominis muscles. Secondary outcomes include functional capacity (SPPB, TUG, 5-time sit-to-stand), handgrip strength, and body composition.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman over 60 years of age, residing in the community, and enrolled in the GPR

Exclusion Criteria:

* Having neuromuscular diseases, recent abdominal surgery, metal implants incompatible with measurements, unstable cardiovascular diseases, or previous participation in another exercise program.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Echo intensity | Baseline and 32 weeks
  Echo intensity (gray scale analysis), using ImageJ software, proposed by the SARCUS consensus and Nutritional Ultrasound ®.
Muscle thickness (mm) | Baseline and 32 weeks
  Linear measurement of the distance between the superficial and deep aponeuroses of a target muscle belly.
Cross-sectional area | Baseline and 32 weeks
  The total area of the muscle (measured in cm^2) in a plane perpendicular to its longitudinal axis
Subcutaneous adipose tissue thickness | Baseline and 32 weeks
  Measurement of the distance between the dermis and the superficial muscle fascia. This variable quantifies the thickness of the fat layer located directly beneath the skin.

SECONDARY OUTCOMES:
Handgrip strength (kg) | Baseline and 32 weeks
  Handgrip strength will be assessed using dynamometry due to its association with various outcomes of aging, being a key component in sarcopenia and frailty. Measurements will be taken using the Hydraulic Jamar device with the subject standing and the elbow flexed at 90º.
Short Physical Performance Battery (SPPB) | Baseline and 32 weeks
  The Short Physical Performance Battery (SPPB) will be used, a quick and objective three-part physical function test with excellent test-retest reliability, predictive validity, and clinical applicability, mainly used for fall risk stratification.
Timed Up and Go (TUG) | Baseline and 32 weeks
  The Timed Up and Go (TUG) test will be used as it is a valid tool for detecting balance deficits, which are associated with an increased risk of falls in older adults.
5-time sit-to-stand (5STS) | Baseline and 32 weeks
  The 5-time sit-to-stand (5STS) test will be used, a functional test serves to assess lower limb strength.
Body Mass Index (BMI) | Baseline and 32 weeks
  alculated as weight in kilograms divided by the square of height in meters (kg/m²). It is used to assess changes in body mass relative to height.
Body Fat Percentage | Baseline and 32 weeks
  Total body fat percentage measured through electrical bioimpedance (BIA) using the TANITA BC-418 device (%).
Abdominal Circumference | Baseline and 32 weeks
  Measured at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest using a flexible tape measure.
Waist-to-Hip Ratio | Baseline and 32 weeks.
  Calculated by dividing the waist circumference by the hip circumference. Used as an indicator of abdominal fat distribution.

OTHER OUTCOMES:
Sociodemographic variables | Baseline and 32 weeks
  Personal data, medical history, presence of comorbidities, use of medications will be collected in a personal interview, and finally, blood pressure will be taken.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Salamanca, Salamanca, Salamanca, Spain